CLINICAL TRIAL: NCT06267274
Title: A Randomized, Double-blind, Parallel-group, Two-arm, Multiple Dose, Multicenter, Bioequivalence Study With Clinical Endpoint Comparing Generic Bimatoprost Ophthalmic Solution 0.01% and LUMIGAN® (Bimatoprost Ophthalmic Solution) 0.01% in the Treatment of Subjects With Chronic Open-angle Glaucoma or Ocular Hypertension in Both Eyes
Brief Title: A Randomized, Double-blind, Parallel-group, Two-arm, Multiple Dose, Multicenter, Bioequivalence Study With Clinical Endpoint in the Treatment of Subjects With Chronic Open-angle Glaucoma or Ocular Hypertension in Both Eyes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: CBCC Global Inc. (Unknown); Amneal EU, Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MW230021
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in such way that ratio of treatment distribution will be nearer to 1:1 between the treatment arms, and within the combined stratification criteria.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimatoprost Ophthalmic Solution, 0.01% (Experimental): Test Product: Bimatoprost Ophthalmic Solution, 0.01%
  Interventions: Drug: Bimatoprost Ophthalmic Solution, 0.01%
- LUMIGAN® (bimatoprost ophthalmic solution) 0.01% (Active Comparator): Reference Product: LUMIGAN® (bimatoprost ophthalmic solution) 0.01%
  Interventions: Drug: LUMIGAN® (bimatoprost ophthalmic solution) 0.01%

INTERVENTIONS:
Drug: Bimatoprost Ophthalmic Solution, 0.01% — 1 drop of ophthalmic solution instill in both eyes every night at 10:00 pm (±1 hours) for 42 days (6 weeks) (± 4 days) as per the randomization schedule.
  Arms: Bimatoprost Ophthalmic Solution, 0.01%
Drug: LUMIGAN® (bimatoprost ophthalmic solution) 0.01% — 1 drop of ophthalmic solution instill in both eyes every night at 10:00 pm (±1 hours) for 42 days (6 weeks) (± 4 days) as per the randomization schedule.
  Arms: LUMIGAN® (bimatoprost ophthalmic solution) 0.01%

SUMMARY:
A randomized, double-blind, parallel-group, two-arm, multiple dose, multicenter, clinical endpoint bioequivalence study

DETAILED DESCRIPTION:
Subjects with chronic open-angle glaucoma or ocular hypertension in both eyes who meet all of the inclusion criteria and none of the exclusion criteria will be identified.

Potential subjects will be screened within 6 weeks prior to administration of the first drop of study drug. They will undergo a washout period of 4 days to 4 weeks (28 days) based on their current medication (if available). Based on stratification criteria, IOP and CCT information available at baseline visit for each subject, the subjects will be randomized in such way that ratio of treatment distribution will be nearer to 1:1 between the treatment arms, and within the combined stratification criteria. The Primary Endpoint is mean difference in the IOP of both eyes between the two treatment groups at 3 time points, i.e., at 00.00 hour, 04.00 hours (4 hours ±1 hour after 00.00 hour), and 08.00 hours (8 hours ±1 hour after 00.00 hour) at Day 14 (Week 2) (± 4 days) and Day 42 (Week 6) (± 4 days) visits.

The Secondary Endpoint: the incidence of all adverse events reported during the study will be summarized by treatment group. Test and reference products will be compared for safety by analyzing nature, severity and frequency of treatment emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to provide voluntary informed consent and to follow protocol requirements.
2. Male or females aged ≥18 years.
3. Subjects with chronic open-angle glaucoma or ocular hypertension in both eyes
4. Subjects requiring treatment of both eyes and able to discontinue the use of all ocular hypotensive medication(s) or switch ocular hypotensive medications and undergo appropriate washout period.
5. Adequate washout period prior to baseline of any ocular hypotensive medications as (to minimize potential risk to subjects due to intraocular pressure (IOP) elevations during the washout period, the Investigator may choose to substitute a parasympathomimetic or carbonic anhydrase inhibitor in place of a sympathomimetic, alpha-agonist, beta-adrenergic blocking agent, or prostaglandin; however, all the subjects must have discontinued their ocular hypotensive medications for the minimum washout period .
6. Baseline (Day 0/hour 0) IOP ≥22 mm Hg and <28 mm Hg in each eye, with difference between the IOP in left and right eyes not being more than 5 mm Hg
7. Subjects' IOP is likely to be controlled with monotherapy as per the Investigator's discretion.
8. Baseline best corrected visual acuity equivalent to Snellen acuity of 20/100 or better in each eye, using a logarithmic visual acuity chart for testing at 10 feet (3 meters).
9. Women of childbearing potential (defined as women physiologically capable of becoming pregnant unless they are using an effective method of contraception during the dosing of the study drug) practicing any of the following acceptable methods of contraception:

   1. Oral or parenteral (injection, patch, or implant) hormonal contraception which has been continuously used for at least 1 month prior to first dose of study medication.
   2. Intrauterine device (IUD) or intrauterine system (IUS)
   3. Double barrier method of contraception (condom and occlusive cap or condom and spermicidal agent)
   4. Male sterilization (at least 6 months prior to screening, should be the sole male partner for that subject)
   5. Female sterilization (surgical bilateral oophorectomy) or tubal ligation at least 6 weeks prior to study participation
   6. Total abstinence; partial abstinence is not acceptable
10. No history of addiction to any recreational drug or drug dependence or alcohol addiction

Exclusion Criteria:

1. Female who are pregnant, lactating or planning a pregnancy.
2. Subjects recently diagnosed with open-angle glaucoma or ocular hypertension and who are treatment naive.
3. Contraindication or known hypersensitivity to Bimatoprost, related class of drugs, or any of the excipients of formulation.
4. Current or history of severe hepatic or renal impairment.
5. Current or history within 2 months prior to baseline of any other significant ocular disease, e.g., corneal edema, uveitis, ocular infection, or ocular trauma in either eye (Note: stable myopia, strabismus, and cataracts as per the Investigator's discretion will be allowed provided that the other inclusion/exclusion criteria are met).
6. Current corneal abnormalities that would prevent accurate IOP readings with Goldmann applanation tonometer.
7. Functionally significant visual field loss in the Investigators' opinion.
8. Subject with corneal grafts.
9. Subject has contraindication to pupil dilation.
10. Use at any time prior to baseline of an intraocular corticosteroid implant.
11. Use of contact lens within 1 week prior to baseline.
12. Use within 2 weeks prior to baseline of 1) a topical ophthalmic corticosteroid or 2) a topical corticosteroid.
13. Use within 1 month prior to baseline of 1) a systemic corticosteroid or 2) high-dose salicylate therapy defined as 325 mg/day and taken on 3 consecutive days.
14. Use within 6 months prior to baseline of intravitreal or subtenon injection of an ophthalmic corticosteroid.
15. Underwent within 6 months prior to baseline any other intraocular surgery (e.g., cataract surgery).
16. Underwent within 12 months prior to baseline any refractive surgery, filtering surgery, or laser surgery for IOP reduction (e.g., laser trabeculoplasty).
17. Amblyopia - only one sighted eye.
18. Subjects with a history of IOP previously uncontrolled on bimatoprost monotherapy.
19. Significant ocular surface findings (e.g., hyperemia or irritation, mild or greater) in either eye found on gross macroscopic or slit lamp examination.
20. Severe retinal disease or other severe ocular pathology, such as glaucomatous damage with a cup/disk ratio greater than 0.8 (not including physiological cupping in the Investigators' opinion) or split fixation.
21. Chronic use of any systemic medication that may affect IOP with less than 3 months stable dosing regimen (i.e., sympathomimetic agents, beta-adrenergic blocking agents, alpha-agonists, alpha-adrenergic blocking agents, calcium channel blockers, angiotensin-converting enzyme inhibitors, etc.)
22. Central Corneal thickness (CCT) <450 microns or >650 microns.
23. Known history or presence of any uncontrolled systemic disease (e.g., cardiovascular disease, hypertension, diabetes mellitus, hepatic impairment, etc.)
24. History of recurrent ocular seasonal allergies within the past 2 years.
25. Any other medical condition or serious intercurrent illness that, in the Investigator's opinion, may make it undesirable for the subject to participate in the study and would limit adherence to the study requirements.
26. Participation in any clinical study within 30 days before the first dose of the study drug.
27. Subjects with known history of positive serology for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV) infection.
28. Subjects with positive urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 00.00 hour, 04.00 hours (4 hours ±1 hour after 00.00 hour), and 08.00 hours (8 hours ±1 hour after 00.00 hour) at Day 14 (Week 2) (± 4 days) and Day 42 (Week 6) (± 4 days) visits
  Mean difference in the IOP of both eyes between the two treatment groups at 3 time points

SECONDARY OUTCOMES:
Secondary Endpoint | AE Monitoring for Safety will be evaluated throughout the study for 6 weeks
  The incidence of all adverse events reported during the study will be summarized by treatment group. Test and reference products will be compared for safety by analyzing nature, severity and frequency of treatment emergent adverse events.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - West Coast Eye Institute, Bakersfield, California
  - Eye Research Foundation, Newport Beach, California
  - Clayton Eye Research, Morrow, Georgia
  - Houston Eye Associates, Houston, Texas

IPD SHARING:
Plan to Share IPD: No